CLINICAL TRIAL: NCT06517173
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Y-3 in Chinese Subjects with Acute Ischemic Stroke
Brief Title: Y-3 for Injection in the Treatment of Acute Ischemic Stroke
Acronym: NUWA-Y3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y-3-LC-04
Record Dates: First submitted 2024-06-28; First posted 2024-07-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Subjects within 48 hours
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Intervention Model Description: This trial is designed as a multicenter, randomized, double-blind, placebo-parallel controlled trial using a multicenter, randomized, double-blind, placebo-parallel controlled trial design. Subjects are randomly assigned in a 1:1 ratio and random number tables are generated using SAS（Statistics Analysis System）software.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Y-3 for injection test group (Experimental): The special solvent Y-3 for injection was extracted with a sterile syringe and injected into a Y-3 lyophilized powder vial for injection. The vial was artificially vibrated until the powder was completely dissolved, and then injected into 250mL 0.9% sodium chloride injection with a sterile syringe for dilution, gently shaken and mixed, and intravenous infusion was performed for 60min±10min. The treatment was performed 10 times for 10 days. The first dose should be completed as soon as possible after randomization; The time from the second dose to the first dose shall not be less than 12h, but not more than 24h+1h. The time interval of each subsequent administration is 24h±1h
  Interventions: Drug: Y-3 for injection
- Placebo control group (Placebo Comparator): The special solvent Y-3 for injection was extracted with a sterile syringe and injected into the lyophilized powder vial of Y-3 simulant for injection. The vial was artificially vibrated until the powder was completely dissolved, and then injected into 250mL 0.9% sodium chloride injection with a sterile syringe for dilution, gently shaken and mixed, and intravenous infusion was performed for 60min±10min. The treatment was performed 10 times for 10 days. The first dose should be completed as soon as possible after randomization; The time from the second dose to the first dose shall not be less than 12h, but not more than 24h+1h. The time interval of each subsequent administration is 24h±1h
  Interventions: Drug: Placebo control group

INTERVENTIONS:
Drug: Y-3 for injection — Qualified subjects were randomly divided into groups in a 1:1 ratio and received continuous treatment with Y-3 injection (40 mg/dose, qd) or placebo control drug. The treatment was performed 10 times for 10 days.
  Arms: Y-3 for injection test group
Drug: Placebo control group — Qualified subjects were randomly divided into groups in a 1:1 ratio and received continuous treatment with Y-3 injection (40 mg/dose, qd) or placebo control drug. The treatment was performed 10 times for 10 days.
  Arms: Placebo control group

SUMMARY:
This trial aims to evaluate the effectiveness and safety of Y-3 for injection in the treatment of patients with acute ischemic stroke within 48 hours of onset

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, parallel, placebo-controlled trial design was adopted, and subjects were randomly assigned to Y-3 for injection group and placebo group in a 1:1 ratio. randomization stratification factors include: onset time (≤12 hours, >12 hours) and research site.

Treatment was continued for 10 days (10 times), and follow-up was conducted until the 90th day from the first dose.

The trial is divided into three phases: screening/baseline phase, treatment phase, and follow-up phase.

Screening/baseline period: After the subjects sign the informed consent form, they enter the screening/baseline period for screening examination.

Treatment period: Qualified subjects are randomly divided into groups in a 1:1 ratio and receive continuous treatment for 10 days (10 times) with Y-3 for injection and placebo respectively. During the treatment period, relevant examinations and evaluations required by the protocol will be carried out; PK blood samples from subjects were collected for population pharmacokinetic analysis.

Follow-up period: Subjects who have completed treatment will enter the follow-up period until the 90th day of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 81 years, male or female;
2. After onset of disease, ischemic stroke meeting the following characteristics: 7≤ NIHSS(National Institutes of Stroke score)≤20 , and the sum of the scores of the item 5 upper limb and item 6 lower limb ≥ 2 points. If patients received thrombolytic therapy, they would be screened and assessed by NIHSS score after thrombolysis;
3. Within 48 hours (inclusive) of onset;
4. Patients who were diagnosed as ischemic stroke according to Key Points in Diagnosis of Various Major Cerebrovascular Diseases 2019 in China and recovered well after the first or last onset of disease (mRS score ≤ 1 point before this episode);
5. The patient or his/her legal representative voluntarily signed informed consent form approved by the Ethics Committee.

Exclusion Criteria:

1. Intracranial hemorrhagic disease by cranial imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.; if it was only oozing, the investigator could determine whether it was suitable for enrollment;
2. Severe disturbance of consciousness: NIHSS score > 1 on item 1a level of consciousness;
3. Transient ischemic attack (TIA);
4. Systolic blood pressure ≥ 220 mmHg or diastolic blood pressure ≥ 120 mmHg after blood pressure control;
5. Previous diagnosis of severe mental disorders and severe dementia;
6. Previously diagnosed with depression or anxiety;
7. Receiving antidepressant or anxiolytic therapy;
8. Have been diagnosed with severe active liver diseases, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc.; or alanine aminotransferase or aspartate aminotransferase > 2.0 × upper limit of normal;
9. Have been diagnosed with severe active renal disease, renal dysfunction; or serum creatinine > 1.5 × upper limit of normal;
10. After this episode, drugs with brain cell protective effect clarified in the package insert have been applied, such as commercially available edaravone,concentrated solution of edaravone and dextranol for injection, nimodipine, ganglioside, citicoline, piracetam, oxiracetam, butylphenyl peptide, human urinary kininogenase (urinary kallidinogenase), cinepazide, rat nerve growth factor, cerebrolysin (brain protein hydrolysate), deproteinized calf serum injection, deproteinized calf blood extract injection, etc.;
11. Thrombectomy or interventional therapy has been applied or planned after this episode;
12. Previous diagnosis of concurrent malignancy and ongoing anti-tumor therapy;
13. Previous diagnosis of severe systemic disease with expected survival times < 90 days;
14. The patient is pregnant, lactating and the patient/patient's partner may become pregnant and plans to become pregnant during the trial;
15. Previously known hypersensitivity to the product or any of its excipients (15-hydroxystearate polyethylene glycol, propylene glycol, mannitol, potassium dihydrogen phosphate, dipotassium hydrogen phosphate trihydrate);
16. History of major surgery within 4 weeks prior to enrollment that impacts neurological score assessed by the investigator or impacts 90-day survival;
17. Participation in another clinical study within 30 days prior to randomization or ongoing participation in another clinical study;
18. Investigator considered inappropriate for participation in this clinical study.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 998 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with Modified Rankin Scale(mRS) score ≤ 1 on the 90th day of treatment | On the 90th day of treatment
  Measure the scores of subjects using the Modified Rankin Scale(mRS) scale.Measure on the 90th day of treatment to evaluate the effectiveness of the medication.The Modified Rankin Scale(mRS) score of this study ranged from 0 to 5. The higher the score, the worse the recovery, and the lower the score, the better the recovery.

SECONDARY OUTCOMES:
Good functional prognosis on the 90th day of treatment | On the 90th day of treatment
  Modified Rankin Scale(mRS) score corrected based on baseline National Institute of Health stroke scale(NIHSS) score. The baseline National Institute of Health stroke scale(NIHSS) score of 4-7 is 0 on the 90 day Modified Rankin Scale(mRS) score; The baseline National Institute of Health stroke scale(NIHSS) score of 8-14 is 0-1 on a 90 day Modified Rankin Scale(mRS) score; The baseline National Institute of Health stroke scale(NIHSS) score is 15-25, with a 90 day Modified Rankin Scale(mRS) score of 0-2. Measure on the 90th day of treatment to evaluate the effectiveness of the medication.
Modified Rankin Scale(mRS) displacement analysis on the 90th day of treatment; | On the 90th day of treatment
  Measure the scores of subjects using the Modified Rankin Scale(mRS). Measure on the 90th day of treatment to evaluate the effectiveness of the medication.The Modified Rankin Scale(mRS) score of this study ranged from 0 to 5. The higher the score, the worse the recovery, and the lower the score, the better the recovery.
The proportion of National Institute of Health stroke scale(NIHSS) scores reduced by ≥ 4 compared to baseline on the 10th and 30th day of treatment; | On the 10th and 30th day of treatment
  Measure the scores of subjects using the National Institute of Health stroke scale(NIHSS). Measure on the 10th and 30th day of treatment to evaluate the effectiveness of the medication.National Institute of Health stroke scale(NIHSS) A larger difference from baseline means a better patient recovery, and a smaller difference means a worse patient recovery.
The proportion of individuals with Barthel Index score ≥ 95 on the 90th day of treatment on the Activities of Daily Living Scale. | On the 90th day of treatment
  Measure the scores of subjects using the Barthel Index scale. Measure on the 90th day of treatment to evaluate the effectiveness of the medication.The total score of the Barthel Index is 100.The higher the Barthel Index scale score, the better the recovery, and the lower the score, the worse the recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] van Horn N, Kniep H, Leischner H, McDonough R, Deb-Chatterji M, Broocks G, Thomalla G, Brekenfeld C, Fiehler J, Hanning U, Flottmann F. Predictors of poor clinical outcome despite complete reperfusion in acute ischemic stroke patients. J Neurointerv Surg. 2021 Jan;13(1):14-18. doi: 10.1136/neurintsurg-2020-015889. Epub 2020 May 15. PMID 32414889
- [Background] Lee SH, Kim BJ, Han MK, Park TH, Lee KB, Lee BC, Yu KH, Oh MS, Cha JK, Kim DH, Nah HW, Lee J, Lee SJ, Kim JG, Park JM, Kang K, Cho YJ, Hong KS, Park HK, Choi JC, Kim JT, Choi K, Kim DE, Ryu WS, Kim WJ, Shin DI, Yeo M, Sohn SI, Hong JH, Lee J, Lee JS, Khatri P, Bae HJ. Futile reperfusion and predicted therapeutic benefits after successful endovascular treatment according to initial stroke severity. BMC Neurol. 2019 Jan 15;19(1):11. doi: 10.1186/s12883-019-1237-2. PMID 30646858
- [Background] Meyer L, Alexandrou M, Leischner H, Flottmann F, Deb-Chatterji M, Abdullayev N, Maus V, Politi M, Roth C, Kastrup A, Thomalla G, Mpotsaris A, Fiehler J, Papanagiotou P. Mechanical thrombectomy in nonagenarians with acute ischemic stroke. J Neurointerv Surg. 2019 Nov;11(11):1091-1094. doi: 10.1136/neurintsurg-2019-014785. Epub 2019 Apr 27. PMID 31030188
- [Background] Chamorro A, Lo EH, Renu A, van Leyen K, Lyden PD. The future of neuroprotection in stroke. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):129-135. doi: 10.1136/jnnp-2020-324283. Epub 2020 Nov 4. PMID 33148815
- [Background] Li J, Zhang L, Xu C, Shen YY, Lin YH, Zhang Y, Wu HY, Chang L, Zhang YD, Chen R, Zhang ZP, Luo CX, Li F, Zhu DY. A pain killer without analgesic tolerance designed by co-targeting PSD-95-nNOS interaction and alpha2-containning GABAARs. Theranostics. 2021 Apr 3;11(12):5970-5985. doi: 10.7150/thno.58364. eCollection 2021. PMID 33897893
- [Background] Li J, Zhang L, Xu C, Lin YH, Zhang Y, Wu HY, Chang L, Zhang YD, Luo CX, Li F, Zhu DY. Prolonged Use of NMDAR Antagonist Develops Analgesic Tolerance in Neuropathic Pain via Nitric Oxide Reduction-Induced GABAergic Disinhibition. Neurotherapeutics. 2020 Jul;17(3):1016-1030. doi: 10.1007/s13311-020-00883-w. PMID 32632774
- [Background] Kaur H, Prakash A, Medhi B. Drug therapy in stroke: from preclinical to clinical studies. Pharmacology. 2013;92(5-6):324-34. doi: 10.1159/000356320. Epub 2013 Dec 12. PMID 24356194
- [Background] Fisher M; Stroke Therapy Academic Industry Roundtable. Recommendations for advancing development of acute stroke therapies: Stroke Therapy Academic Industry Roundtable 3. Stroke. 2003 Jun;34(6):1539-46. doi: 10.1161/01.STR.0000072983.64326.53. Epub 2003 May 15. PMID 12750546
- [Background] Hackett ML, Kohler S, O'Brien JT, Mead GE. Neuropsychiatric outcomes of stroke. Lancet Neurol. 2014 May;13(5):525-34. doi: 10.1016/S1474-4422(14)70016-X. Epub 2014 Mar 28. PMID 24685278
- [Background] Ferro JM, Caeiro L, Figueira ML. Neuropsychiatric sequelae of stroke. Nat Rev Neurol. 2016 May;12(5):269-80. doi: 10.1038/nrneurol.2016.46. Epub 2016 Apr 11. PMID 27063107
- [Background] Murrough JW, Abdallah CG, Mathew SJ. Targeting glutamate signalling in depression: progress and prospects. Nat Rev Drug Discov. 2017 Jul;16(7):472-486. doi: 10.1038/nrd.2017.16. Epub 2017 Mar 17. PMID 28303025
- [Background] Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011 Apr;16(4):383-406. doi: 10.1038/mp.2010.120. Epub 2010 Nov 16. PMID 21079608
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] Griebel G, Holmes A. 50 years of hurdles and hope in anxiolytic drug discovery. Nat Rev Drug Discov. 2013 Sep;12(9):667-87. doi: 10.1038/nrd4075. PMID 23989795
- [Background] Shabel SJ, Proulx CD, Piriz J, Malinow R. Mood regulation. GABA/glutamate co-release controls habenula output and is modified by antidepressant treatment. Science. 2014 Sep 19;345(6203):1494-8. doi: 10.1126/science.1250469. Epub 2014 Sep 18. PMID 25237099
- [Background] Li YF. A hypothesis of monoamine (5-HT) - Glutamate/GABA long neural circuit: Aiming for fast-onset antidepressant discovery. Pharmacol Ther. 2020 Apr;208:107494. doi: 10.1016/j.pharmthera.2020.107494. Epub 2020 Jan 25. PMID 31991195
- [Background] Gould TD, Zarate CA Jr, Thompson SM. Molecular Pharmacology and Neurobiology of Rapid-Acting Antidepressants. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:213-236. doi: 10.1146/annurev-pharmtox-010617-052811. Epub 2018 Oct 8. PMID 30296896
- [Background] Zhou L, Li F, Xu HB, Luo CX, Wu HY, Zhu MM, Lu W, Ji X, Zhou QG, Zhu DY. Treatment of cerebral ischemia by disrupting ischemia-induced interaction of nNOS with PSD-95. Nat Med. 2010 Dec;16(12):1439-43. doi: 10.1038/nm.2245. Epub 2010 Nov 21. PMID 21102461
- [Background] Luo CX, Lin YH, Qian XD, Tang Y, Zhou HH, Jin X, Ni HY, Zhang FY, Qin C, Li F, Zhang Y, Wu HY, Chang L, Zhu DY. Interaction of nNOS with PSD-95 negatively controls regenerative repair after stroke. J Neurosci. 2014 Oct 1;34(40):13535-48. doi: 10.1523/JNEUROSCI.1305-14.2014. PMID 25274829
- [Derived] Li S, Wang X, Feng B, Li H, Wang Y. Loberamisal for Acute Ischaemic Stroke (LAIS): a multicentre, randomised, double-blind, parallel, placebo-controlled phase III clinical trial. Stroke Vasc Neurol. 2025 Dec 4:svn-2025-004582. doi: 10.1136/svn-2025-004582. Online ahead of print. PMID 41344725